CLINICAL TRIAL: NCT03398811
Title: Predictors of Abnormal Uterine Bleeding in Progestin-only Contraceptives Users
Brief Title: Abnormal Uterine Bleeding and Progestin-only Contraceptives
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Other Study IDs: POCU
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel; Desogestrel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I "the depot medroxy-progesterone acetate group": where they will use Depot Medroxyprogesterone Acetate 150 mg injection every 3 month,
  Interventions: Drug: Depot medroxy-progesterone acetate
- Group II "Implanon group": where they will have Implanon (etonogestrel implant) 68 mg implant
  Interventions: Drug: Etonogestrel
- group III (cerazette group): where they are using Cerazette pills (desogestrel 75 µg l) one pill every day for 28 days without pill-free interval.
  Interventions: Drug: Desogestrel 75 µg

INTERVENTIONS:
Drug: Depot medroxy-progesterone acetate — Injection every 3 months
  Groups: Group I "the depot medroxy-progesterone acetate group"
Drug: Etonogestrel — 68 mg implant
  Groups: Group II "Implanon group"
Drug: Desogestrel 75 µg — one pill every day for 28 days without pill-free interval.
  Groups: group III (cerazette group)

SUMMARY:
The use of progestin-only methods of contraception has been increased obviously and progressively over the world in the last few years. Progestin-only contraception is an option for women in whom an estrogen-containing contraceptive is either contraindicated or causes additional health concerns.

Progestogen-only pills are contraceptive pills that contain only synthetic progestogens (progestins) and do not contain estrogen . The progestin-only pill is recommended over regular birth control pills for women who are breastfeeding because the mini-pill does not affect milk production.

The most common progestin-only method used is the injectable depot medroxy-progesterone acetate which had been approved by Food and Drug Administration since 1992 . depot medroxy-progesterone acetate provides reliable, private, long-acting (three months) and reversible contraception. Users of depot medroxy-progesterone acetate don't need daily taking as well as it doesn't affect the intercourse by any mean.

The etonogestrel implant (Implanon) is a single-rod progestin contraceptive method placed subdermally in the inner aspect of upper non dependant arm for three years. Much evidence supports the safety, efficacy, reversibility and acceptability of this contraceptive method.

A common reason women choose to discontinue progestin-only contraception is dissatisfaction with its effects on uterine bleeding which occurs in a significant number of users. Information revealed from many clinical trials shows that abnormal uterine bleeding with progestin-only contraception ranging from 10 to 25 % at first year of use.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18-40 years.
2. Women with more than 12 month postpartum.
3. Women who had normal menstrual pattern (cycle from 21 - 35 days with a same cycle length variation of no more than 5 days, bleeding days from 2-7 days and number of sanitary pads not more than 3 pads without blood clots or flooding of blood).
4. Women wanted to use DMPA, etonogestrel subdermal implant or POPs only for pregnancy prevention for at least 1 year.

Exclusion Criteria:

1. Women on any anticoagulant therapy.
2. Women who had a history of uterine, cervical or ovarian pathology.
3. Women who had uterine bleeding disturbance (including amenorrhea) before recruitment.
4. Women received DMPA injection within the previous 9 months except they had three spontaneous regular menstrual cycles.
5. Severely anemic women (hemoglobin < 8gm/dl).
6. Women with any contraindications for POCs following the WHO eligibility (Altshuler AL et al., 2015).
7. Women refused to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women who requested DMPA, etonogestrel subdermal implant or POPs for pregnancy prevention.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Number of women developed vaginal bleeding | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided